CLINICAL TRIAL: NCT04652310
Title: Long vs Extended-short Nail When Treating Proximal Femur Fractures - An RCT-study Examining Differences in Functional and Surgical Outcomes
Brief Title: Long vs Extended-short Nail When Treating Proximal Femur Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REK 2019/125
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Hip Fractures
Keywords: intramedullary nailing; TFNA
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended-Short Nail (Active Comparator): Implantation of TFNA extended-short nail (235 mm)
  Interventions: Device: TFNA extended-short nail (235 mm)
- Long nail (Active Comparator): Implantation of TFNA long nail (260-480 mm)
  Interventions: Device: TFNA long nail (260-480mm)

INTERVENTIONS:
Device: TFNA extended-short nail (235 mm) — The extended short version of the TFN-advanced proximal femoral nailing system (TFNA)
  Other Names: TFN-advanced proximal femoral nailing system (TFNA) 235 mm
  Arms: Extended-Short Nail
Device: TFNA long nail (260-480mm) — The long version of the TFN-advanced proximal femoral nailing system (TFNA)
  Other Names: TFN-advanced proximal femoral nailing system (TFNA) 260-480mm
  Arms: Long nail

SUMMARY:
Fractures of the upper part of the femur may be treated with intramedullary nails. There are different designs to choose from. The intention of this RCT is to compare two nails with some of the same properties, but with different lengths. Usually, it is the surgeon who decides which nail to be used. The literature indicates that there is a lack of good evidence in the decision-making, and that the choice often depends on personal preferences and experience of the surgeon. Therefore, the investigators want to compare whether one of the nails has a better outcome than the other, and in that way be able to give some clearer guidelines for treatment. Patients will be randomized into two groups, one receiving a long nail and one receiving an extended-short nail and compare surgical and functional outcomes. Information from the operation and subsequent check-ups will be analysed. The hypothesis is that the extended-short nail can reduce operating time, bleeding, fluoroscopy time and give equal or better functional outcome, without increasing reoperation rates or mortality.

DETAILED DESCRIPTION:
Background Intramedullary nails have in recent years become the preferred technique compared to DHS when treating proximal femur fractures. A Norwegian RCT has showed the same frequency of postoperative pain, functional outcome and rate of reoperations comparing the two techniques. Nails are usually provided in a long and short model. Deciding which nail length to use is highly discussed, and often a long nail is preferred, because it gives a theoretically more stable and secure fixation of the femur. There are, however many advantages of using a short nail. It is less time consuming as there is no need for reaming, securing the long nail distally requires more fluoroscopy time, and distal locking of the long nail has also been shown to increase the risk of perioperative fractures. Perioperative bleeding and postoperative blood transfusions are reduced when using a short nail, and a long nail may also give more pain distally around the thigh and around the knee owing to cortical impingement. Finally, the long nail is more expensive compared to short models. There is a perception in the orthopedic society that there's a higher risk of periprosthetic fractures with short nails, but the latest generations of nails have improved this problem. Most studies report no difference in periprostetic fractures between long and short nails. Recently, new extended-short versions of medullary nails are being produced. The extended-short nail combines the mechanical properties seen in a long nail and the surgical simplicity of a short nail. This new nail type may replace the use of several long nails being placed just to be on the safe side, and thus reduce operating time, bleeding and postoperative pain associated with a long nail. Biomechanical studies have showed that the mechanical properties of long and extended-short nails are predominantly comparable, but to our knowledge no clinical studies comparing the extended-short and long nails have been performed to date. The advantages of an extended-short nail are potentially great, which makes it important to clarify which opportunities there are to benefit from this type of nail for certain types of fractures, both in the interest of the patient as well as the economic healthcare perspective.

Purpose In a well-defined population of patients with proximal femur fractures within a certain anatomical area the aim is to compare the extended-short nail with the long nail, to evaluate differences in functional and surgical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Intertrochanteric, pertrochanteric or subtrochanteric fractures
* Distal fracture limit within 4 cm below the trochanter minor
* Intramedullary nailing with TFNA-nail is indicated
* Patient is fit for surgery.

Exclusion Criteria:

* AO 31-A3 fractures (revers oblique fractures)
* Cognitively impaired patients who themselves cannot understand the study information and give informed consent, and do not have a next of kin or legal guardian who can give consent on their behalf.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Difference in Short Physical Performance Battery (SPPB)-score | At 3 months and 1 year
  Short Physical Performance Battery (SPPB)-score, ranges from 0-12, 12 is the best indicating a good physical function.

SECONDARY OUTCOMES:
Difference in Operation time | Surgery date
  Operation time in minutes
Difference in Blood loss | Surgery date
  Blood loss during surgery
Difference in Harris Hip score | 3 months and 1 year
  Harris Hip score, ranges from 0-100, 100 is the best score, a high score indicates good physical function.
Difference in EQ5D-5L (EuroQoL 5L - health-related quality of life) | 3 months and 1 year
  EQ5D-5L (EuroQoL 5L - health-related quality of life)measures health status terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three-level (EQ-5D-3L) or five-level (EQ-5D-5L) scale
Difference in Transfusion after surgery | 2 weeks after surgery
  Need for transfusion of blood products after surgery
Difference in Fluoroscopy time | Surgery date
  Fluoroscopy time during surgery
Difference in Postoperative complications | Minimally 1 year
  Any postoperative complications
Difference in Mortality | Minimally 1 year
  Mortality after surgery
Difference in Reoperations | Minimally 1 year
  Reoperations of any kind

CONTACTS AND LOCATIONS:
Overall Officials: Heidi B Dyrop, MD, PHD, Principal Investigator — Orthopedic Dpt, Kongsberg Hospital, Vestre Viken HF
Locations (2):
- Norway (2):
  - Drammen Hospital, Vestre Viken HF, Drammen
  - Kongsberg hospital, Vestre Viken HF, Kongsberg

IPD SHARING:
Plan to Share IPD: No